CLINICAL TRIAL: NCT05824702
Title: A Social Network Approach for Improving Medication Assisted Treatment and HIV
Brief Title: A Social Network Approach for Improving Medication Assisted Treatment and HIV Prevention and Medical Care Among People Who Inject Drugs in Ukraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Ukrainian Institute on Public Health Policy (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA051316 (NIH); IRB00024358 (Other: JHSPH IRB); R34DA051316 (NIH)
Record Dates: First submitted 2023-04-05; First posted 2023-04-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: HIV
Keywords: HIV; Drug Treatment

STUDY DESIGN:
Intervention Model Description: A pilot randomized clinical trial of behavioral intervention
Who Masked: Participant
Masking Description: Participants are not aware of the other condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Peer education and network support (Experimental): The intervention sessions will consist of 6 group sessions including 1) Introduction to Peer Educator role and peer Communication skills, 2) HIV and drug treatments, 3) using a decision balance tool with network members for drug treatment, 4) Promoting HIV prevention and medical care & using text messages as peer educators for promoting MAT and HIV prevention and care, 5) Preventing and responding to relapse, and 6) HIV care retention and medication adherence.
  Interventions: Behavioral: Peer education & communications
- comparison: Standard of care of health education (Active Comparator): The comparison condition will include 5 group sessions focused on: 1) retention in MAT by addressing the myths about MAT; 2) information to MAT clients on finding local MAT and other health services in areas where they migrate; 3) importance of HIV prevention (including PreP) and HIV treatment including adherence to HIV; 4) harm reduction, safe drug use, overdose prevention and first aid in case of overdose; 5) addressing Hepatitis C, chronic conditions and mental health issues by emphasizing the importance of timely addressing these health problems and providing information on available local and national services.
  Interventions: Behavioral: Standard of care educational

INTERVENTIONS:
Behavioral: Peer education & communications — The intervention trains peer educators to promote medication-assisted drug treatment among peer who inject drugs and are living with HIV.
  Arms: Experimental: Peer education and network support
Behavioral: Standard of care educational — This is an educational equal attention control group
  Arms: comparison: Standard of care of health education

SUMMARY:
The aim of this study is to pilot a peer education for people on medication assisted treatment (MAT). People on MAT will be trained to be peer educators and provide outreach to the educators social network members who inject drugs, some of whom will be HIV positive.

DETAILED DESCRIPTION:
The, goal of the intervention is to increase medication assisted treatment (MAT) uptake and retention in order to enhance as well as HIV medical care and antiretroviral therapy (ART) adherence among those social network members who use drugs and those living with HIV who use drugs. The project will quantitatively and qualitatively assess barriers to MAT and ART uptake and adherence, while using peer educators to promote MAT and ART among their network members. Finally, the project aims to determine the effect size for guiding the planning of larger intervention and the feasibility and acceptability of this intervention for HIV prevention and improvement in HIV-related health outcomes among people living with HIV who inject drugs (PLWH PWID). The intervention will be deployed in Ukraine, a setting with high HIV incidence rates among PWID, low levels of viral suppression among HIV positive PWID, and low rates of MAT uptake.

ELIGIBILITY:
Inclusion Criteria:

* On methadone for at least 1 year and rated by the staff as low risk for relapse
* Report at least 1 drug network member living with HIV, not on methadone, and seen weekly
* Willing to talk with drug users in their network about medication for drug dependence and accompany them to methadone clinic

Exclusion Criteria:

• Persons that are currently psychotic, suicidal, or cognitively impaired such that they cannot provide informed consent will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Enrolled in drug treatment | 3 months
  Enrollment in drug treatment among social network members living with HIV

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Latkin, Ph.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Ukrainian Institute on Public Health Policy, Kiev, Kyiv Oblast, Ukraine